CLINICAL TRIAL: NCT01509859
Title: Prospective Randomized Trial Comparing the Weight Bearing After Fixation of Proximal Femur Fractures With Two Different Proximal Intramedullary Devices
Brief Title: Comparing Weight Bearing After Intramedullary Fixation Devices for the Proximal Femur Fracture
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, yona kosashvili, senior surgeon, joint arthroplasty unit, orthopedic department, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0333-11-RMC
Record Dates: First submitted 2012-01-05; First posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Closed Comminuted Oblique Intertrochanteric Fracture of Neck of Right Femur; Closed Comminuted Oblique Intertrochanteric Fracture of Neck of Left Femur
Keywords: proximal femur nail; pfna; intertan; weight bearing; pertrochanteric fracture; femur neck fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PFNA (Active Comparator): these patients will be treated with "synthes" PFNA" device
  Interventions: Device: PFNA proximal femur nail device (Synthes)
- INTERTAN (Active Comparator): these patients will be treated with Smith&Nephew "INTERTAN" device
  Interventions: Device: INTERTAN proximal femur nail device (Smith&Nephew)

INTERVENTIONS:
Device: PFNA proximal femur nail device (Synthes) — synthes "PFNA" proximal femur nail device
  Arms: PFNA
Device: INTERTAN proximal femur nail device (Smith&Nephew) — Smith&Nephew "INTERTAN" proximal femur nail device
  Arms: INTERTAN

SUMMARY:
The purpose of the study is to Compare the stability of the fracture and pain after surgery by measuring the stride length and weight bearing on the operated leg. This study will compare these parameters between two different proximal femur nails used for fixing hip fractures.

DETAILED DESCRIPTION:
Fractures of the proximal femur and hip are relatively common injuries in adults.

According to the Evans and the AO Classification systems, the fracture can be described as stable after reduction or not according to the direction of the fracture lines and the comminution of the medial cortex or the lateral wall of the proximal femur.

Biomechanically, nails allow for stable anatomical fixation of more comminuted fractures without shortening the abductor moment arm or changing the proximal femoral anatomy. These devices provide fracture stability by virtue of allowing the lateral aspect of the head and neck to come to rest against the nail in the medullary canal.

For fractures with comminuted medial cortex or involvement of the lateral cortex (AO 2.2 - AO 3.3) it is advisable to fixate with a more stable fixation device such as intramedullary proximal femur nail Several intramedullary devices are currently in use for the treatment of the intertrochanteric fractures. In our institution, for the unstable fracture we use either one of the intramedullary devices manufactured by Synthes (Proximal femoral nail - anti-rotation = PFNA) or by Smith&Nephew (Trochanteric Antegrade Nail = InterTan).

Each of these nails allow compression over the Nail\Blade with the intramedullary stability.

There are 3 main complications in the treatment of intramedullary devices : (1) varus collapse of the head/neck, (2) uncontrolled shortening of the neck, and (3)femoral shaft fractures at the tip of the nail The InterTan, unlike other devices, allows for immediate intraoperative compression of the principal fracture fragments through linear compression combined with rotational stability secondary to its unique geometry and mechanism of action.

The mechanical stability of the fracture after the fixation is reflected by the weight bearing the patient can hold . In order to find weather there is a mechanical difference between the two devices we would like to perform a test measuring the weight bearing after fixation of intertrochanteric fractures comparing the pain and impression of mechanical stability in the two devices.

The method to test the amount of weight bearing would be using the "SmartStep gait system" TM (Andante Medical Devices Ltd), an innovative biofeedback and monitoring system that records and analyzes key gait parameters and provides instantaneous and accurate audio and visual feedback.

ELIGIBILITY:
Inclusion Criteria:

* pertrochanteric fracture ao 2.2 and above
* ambulatory patient, without support prior to the fall
* minor trauma mechanism
* without other injuries
* operated 3 days from the injury

Exclusion Criteria:

* dementia
* s/p hip or knee arthroplasty
* known osteoarthritis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

SECONDARY OUTCOMES:
complication | the patients will be measured during the hospital stay (average of 1 week) and at 6 weeks after surgery
  complication as non union, infection, cut-out will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: yona kosashvili, MD, Principal Investigator — Rabin Medical Center; eliezer sidon, MD, Study Director — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Zlowodzki M, Zelle BA, Cole PA, Jeray K, McKee MD; Evidence-Based Orthopaedic Trauma Working Group. Treatment of acute midshaft clavicle fractures: systematic review of 2144 fractures: on behalf of the Evidence-Based Orthopaedic Trauma Working Group. J Orthop Trauma. 2005 Aug;19(7):504-7. doi: 10.1097/01.bot.0000172287.44278.ef. PMID 16056089
- [Background] Sadowski C, Lubbeke A, Saudan M, Riand N, Stern R, Hoffmeyer P. Treatment of reverse oblique and transverse intertrochanteric fractures with use of an intramedullary nail or a 95 degrees screw-plate: a prospective, randomized study. J Bone Joint Surg Am. 2002 Mar;84(3):372-81. PMID 11886906
- [Background] Cummings SR, Rubin SM, Black D. The future of hip fractures in the United States. Numbers, costs, and potential effects of postmenopausal estrogen. Clin Orthop Relat Res. 1990 Mar;(252):163-6. PMID 2302881
- [Background] Gullberg B, Duppe H, Nilsson B, Redlund-Johnell I, Sernbo I, Obrant K, Johnell O. Incidence of hip fractures in Malmo, Sweden (1950-1991). Bone. 1993;14 Suppl 1:S23-9. doi: 10.1016/8756-3282(93)90345-b. PMID 8110516
- [Background] Williams WW, Parker BC. Complications associated with the use of the gamma nail. Injury. 1992;23(5):291-2. doi: 10.1016/0020-1383(92)90169-s. PMID 1644453
- [Background] Koval KJ, Sala DA, Kummer FJ, Zuckerman JD. Postoperative weight-bearing after a fracture of the femoral neck or an intertrochanteric fracture. J Bone Joint Surg Am. 1998 Mar;80(3):352-6. doi: 10.2106/00004623-199803000-00007. PMID 9531202